CLINICAL TRIAL: NCT00627497
Title: A Prospective, Randomized, Controlled Pivotal Clinical Investigation of DIAM™ Spinal Stabilization System in Patients With Degenerative Lumbar Spinal Stenosis.
Brief Title: DIAM™ Spinal Stabilization System vs. Decompression, Formerly vs. Posterolateral Fusion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow patient recruitment
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05-05 and P07-03
Record Dates: First submitted 2008-02-21; First posted 2008-03-03 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2012-04

CONDITIONS: Degenerative Lumbar Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DIAM Group1 (Experimental)
  Interventions: Device: DIAM Spinal Stabilization
- Single-Level Posterior Decompression (Active Comparator)
  Interventions: Procedure: Single-Level Posterior Decompression
- DIAM Group2 (Experimental)
  Interventions: Device: DIAM Spinal Stabilization
- Posterolateral Interbody Fusion (Active Comparator)
  Interventions: Device: Fusion

INTERVENTIONS:
Procedure: Single-Level Posterior Decompression — The single level posterior decompression is a posterior surgical procedure.
  Arms: Single-Level Posterior Decompression
Device: DIAM Spinal Stabilization — The DIAM Spinal Stabilization System is a spacer that is implanted between adjoining spinous processes using a posterior surgical approach.
  Arms: DIAM Group1
Device: DIAM Spinal Stabilization — The DIAM Spinal Stabilization System is a spacer that is implanted between adjoining spinous processes using a posterior surgical approach
  Arms: DIAM Group2
Device: Fusion — Posterolateral Interbody Fusion
  Arms: Posterolateral Interbody Fusion

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness of the DIAM Spinal Stabilization System as a method of treating patients with symptoms of degenerative lumbar spinal stenosis at a single level from L2 to L5.

DETAILED DESCRIPTION:
This pivotal clinical trial is being conducted to evaluate the DIAM Spinal Stabilization System for the treatment of single-level degenerative lumbar spinal stenosis from L2 to L5. The implant under investigation in this clinical trial is the DIAM Spinal Stabilization System. And following a decompression procedure, the device will be implanted using a posterior surgical approach. Patients in the control group will receive a lumbar decompression.

ELIGIBILITY:
Inclusion Criteria:

* Has a symptom complex consisting of back, buttock, or groin pain (excluding symptomatic coxarthrosis) with leg pain typical of intermittent neurogenic claudication, which is defined as leg(usually calf) discomfort, pain, numbness, paresthesias, weakness, or fatigue aggravated by standing or walking and is only relieved with resting in flexed lumbar spine position
* Leg pain score ≥ 8 and back pain score ≥ 6 based on the Preop Back/ Leg Pain CRF.

Leg pain score must be ≥ back pain score

* Narrowing of the lumbar spinal canal and/or intervertebral foramen at L2-L3, L3-L4, L4-L5 as indicated by MRI, with other MRI findings typical of spinal stenosis, such as trefoil canal shape; hypertrophy, thickening, buckling, or infolding of the ligamentum flavum; hypertrophied facet joints or facet joint capsule; annular bulging; or lateral (subarticular) stenosis.
* Must sit for at least 30 min without severe pain
* Must walk at least 100 ft unassisted
* 35 yrs of age, inclusive
* Preoperative Oswestry score ≥ 40
* Child-bearing potential, pt is not pregnant or nursing and agrees not to become pregnant during study period
* Treated non-operatively for a pd of at least 6 mos
* Willing and able to comply with study plan and able to understand and sign Pt ICF

Exclusion Criteria:

* Disease state which requires destabilizing decompression
* Axial back pain with no pain in leg, buttock, or groin
* Baseline strength grade of 0 (total paralysis), 1 (palpable or visible contraction), or 2 (active movement, gravity,eliminated) in any lower extremity motor group as noted on Neuro Status CRF
* Segmental kyphosis >0° at indicated level
* Cauda equina syndrome
* Compression of nerve roots that causes neurogenic bowel, bladder dysfunction
* Prior surgical procedure at involved or adjacent levels
* Diagnosed with significant peripheral neuropathy
* Significant vascular disease causing vascular claudication
* Requires tx of spinal stenosis at more than 1 lumbar level
* Significant lumbar instability, defined as > 3mm translation on flexion/extension radiographs
* Has > 3mm fixed spondylolisthesis at affected level
* BMI ≥ 40
* Sustained vertebral or hip fracture within last year
* Has the following (if "Yes" to any risk below, a lumbar spine DEXA Scan is required for eligibility)

  1. Previous diagnosis of osteoporosis, osteopenia, or osteomalacia
  2. Postmenopausal Non-Black female over age of 60 who weighs ≤ 140 lbs
  3. Postmenopausal female who has sustained a non traumatic hip, spine or wrist fracture
  4. Male over age of 60 who has sustained non-traumatic hip or spine fracture
* If level of DEXA T-score is -1.0 or lower pt is excluded from study
* Lumbar scoliosis with Cobb angle of > 15°
* Documented allergy to silicone, polyethylene, titanium or latex
* Overt or active bacterial infection, local, systemic, and/or potential for bacteremia
* Alcohol and/or drug abuser
* Received tx with investigational therapy (device and/or pharmaceutical) within 30 days prior to entering study or such tx is planned during the 24 mos following enrollment in study
* Suppressed immune system or has taken steroids at any dose daily for more than 1 mon within the last yr
* Presence of active malignancy or prior history of malignancy except for basal cell carcinoma of the skin
* History of any endocrine or metabolic disorder known to affect osteogenesis
* Chronic or acute renal and/or hepatic failure or prior history of renal and/or hepatic parenchymal disease
* History of autoimmune disease
* Disease which precludes accurate clinical evaluation of safety and effectiveness of txs in this study
* Congenital or iatrogenic posterior element insufficiency
* Moderate to advance spondylosis or pts who demonstrate advanced degenerative changes. Such advanced degenerative changes are characterized by 1 or combination of the following a Bridging osteophytes; b Reduction or absence of motion; c Collapse of the intervertebral disc space of > 50% of its normal ht
* Mentally incompetent
* Waddell Signs of Inorganic Behavior score of ≥ 3
* Prisoner

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Fremont, California
  - Jacksonville, Florida
  - Melbourne, Florida
  - Temple Terrace, Florida
  - Columbus, Georgia
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Winston-Salem, North Carolina
  - Chattanooga, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- DIAM Group1; DIAM Group2: Patients in this group were implanted DIAM Spinal Stabilization System using a posterior surgical approach.
- Single-Level Posterior Decompression: Patients in this group received a single-level posterior lumbar decompression
- Posterolateral Interbody Fusion: Patients in this group received a posterolateral interbody fusion.
Period: Overall Study
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Started | 14 | 12 | 4 | 2
Completed | 13 | 11 | 4 | 2
Not Completed | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion | Total
Number analyzed (Participants) | 14 | 12 | 4 | 2 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (8.3) | 54.8 (9.7) | 47.8 (16.1) | 54.5 (7.8) | 54.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 2 | 2 | 14
  Male | 12 | 4 | 2 | 0 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 11 | 12 | 4 | 2 | 29
  Black | 2 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Hispanic | 1 | 0 | 0 | 0 | 1
  other | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: in.] | 70.1 (3.2) | 66.9 (4.4) | 69.3 (4.3) | 65.5 (0.7) | 68.5 (4.0)
Weight [Mean (Standard Deviation); unit: lbs] | 209.9 (42.0) | 187.2 (36.2) | 194.0 (43.3) | 144.5 (36.1) | 195.3 (41.5)
Oswestry Disability Index (ODI) Score [Mean (Standard Deviation); unit: Scores on a scale] — The Oswestry Disability Index (ODI) Questionnaire was used to assess patient pain and ability to function. The ODI score ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
  Scores on a scale | 52.6 (9.7) | 49.6 (8.4) | 52.0 (10.7) | 44.0 (2.8) | 50.9 (9.0)
General Health Status [Mean (Standard Deviation); unit: Scores on a scale] — The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results are summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS and MCS is between 0 and 100, with higher scores denoting better quality of life. No overall score (SF-36) was reported.
  Scores on a scale
    Physical Component Summary (SF- 36 PCS) | 27.0 (7.9) | 26.6 (4.7) | 27.0 (3.7) | 24.0 (1.5) | 26.7 (6.0)
    Mental Component Summary (SF-36 MCS) | 51.7 (9.2) | 49.7 (10.5) | 46.0 (10.7) | 59.9 (4.2) | 50.7 (9.8)
Pain Status [Mean (Standard Deviation); unit: Scores on a scale] — Numerical rating scales are used to evaluate back pain and leg pain intensity and frequency. Patients will rate their pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients will record their back pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." A patient's total pain score will be the sum of pain intensity and frequency scores (0 min, 20 max).
  Scores on a scale
    Back Pain Score (0-20) | 14.1 (3.1) | 12.0 (3.5) | 15.0 (3.4) | 11.5 (0.7) | 13.3 (3.3)
    Leg Pain Score (0-20) | 17.2 (1.5) | 17.1 (1.7) | 16.8 (3.9) | 16.0 (4.2) | 17.0 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Overall Success
Description: Rate of overall success is reported as the percentage of partipants who met all of the following criteria:
  1. Pain/disability (ODI) success:(Success of ODI is defined as pain/disability improvement according to the definition: Pre-treatment Score - Post-treatment Score ≥ 15);
  2. Neurological success (Neurological success is defined as maintenance or improvement in sections of motor, sensory, reflex, and straight leg raise for the time period evaluated);
  3. No serious adverse event classified as "surgical treatment associated";
  4. No additional surgical procedure classified as "failure."
Time Frame: 24 months after operation
Measure: Number; unit: percentage of patients
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 11 | 4 | 2
percentage of patients | 53.8 | 27.3 | 100.0 | 50.0

2. Secondary Outcome: Oswestry Disability Index (ODI) Score
Description: The self-administered Oswestry Disability Index (ODI) Questionnaire was used to assess patient pain and ability to function. The ODI scale ranges from 0-100. The best score is 0 (no disability) and worst is 100 (maximum disability).
Time Frame: 24 month after operation
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
Scores on a scale
  Oswestry Disability Index (ODI) Score at baseline | 52.6 (9.7) | 49.6 (8.4) | 52.0 (10.7) | 44.0 (2.8)
  Oswestry Disability Index (ODI) Score at 24 month | 15.6 (16.1) | 13.3 (15.6) | 14.1 (10.9) | 20.0 (22.6)
  Change of ODI Score at 24 month from baseline | -37.6 (19.0) | -36.4 (14.6) | -37.9 (11.4) | -24.0 (19.8)

3. Secondary Outcome: Success Rate of Oswestry Diability Index Scores
Description: Success rate of Oswestry Diability Index Scores is reported as the percentage of participants who met: Pre-treatment Score - Post-treatment Score ≥ 15.
Time Frame: 24 month after operation
Measure: Number; unit: percentage of participants
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
percentage of participants | 84.6 | 100.0 | 100.0 | 50.0

4. Secondary Outcome: Success Rate of Neurological Status
Description: Success rate of neurological status is reported as the percentage of participants who met neurological success defined as maintenance or improvement in all sections (motor, sensory, reflex, and straight leg raising) for the time period evaluated. In order for a section to be considered a success, each element in the section must remain the same or improve from the time of the preoperative evaluation to the time period evaluated.
Time Frame: 24 month after operation
Measure: Number; unit: percentage of particpants
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
percentage of particpants | 61.5 | 37.5 | 100.0 | 100.0

5. Secondary Outcome: Back Pain
Description: Numerical rating scales are used to evaluate back pain intensity and frequency. Patients will rate their pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients will record their back pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." A patient's total pain score will be the sum of pain intensity and frequency scores (0 min, 20 max).
Time Frame: 24 month after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
units on a scale
  Back Pain Score at baseline | 14.1 (3.1) | 12.0 (3.5) | 15.0 (3.4) | 11.5 (0.7)
  Back Pain Score at 24 month | 5.4 (5.7) | 6.9 (7.2) | 6.5 (4.7) | 5.0 (2.8)
  Pain Score change at 21 month from baseline | -8.9 (6.2) | -5.9 (5.2) | -8.5 (5.4) | -6.5 (3.5)

6. Secondary Outcome: Back Pain Success Rate
Description: Back pain success rate is reported as the percentage of participants whose back pain improvement met: (Pre Score - Post Score)/ Pre Score > 20%.
Time Frame: 24 month after operation
Measure: Number; unit: percentage of participants
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
percentage of participants | 76.9 | 75.0 | 100.0 | 100.0

7. Secondary Outcome: Leg Pain
Description: Numerical rating scales are used to evaluate leg intensity and frequency. Patients will rate their pain intensity on a scale from 0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be." Similarly, patients will record their back pain frequency on a scale from 0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time." A patient's total pain score will be the sum of pain intensity and frequency scores (0 min, 20 max).
Time Frame: 24 month after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
units on a scale
  Leg Pain at baseline | 17.2 (1.5) | 17.1 (1.7) | 16.8 (3.9) | 16.0 (4.2)
  Leg pain at 24 month | 5.7 (6.5) | 8.5 (9.2) | 2.0 (2.7) | 3.0 (4.2)
  Pain Score change at 24 month from baseline | -11.7 (6.5) | -8.8 (9.0) | -14.8 (6.6) | -13.0 (0.0)

8. Secondary Outcome: Leg Pain Success Rate
Description: Leg pain success rate is reported as the percentage of participants whose leg pain improvement met: (Pre Score - Post Score)/ Pre Score > 20%.
Time Frame: 24 month after operation
Measure: Number; unit: percentage of participant
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
percentage of participant | 84.6 | 62.5 | 100.0 | 100.0

9. Secondary Outcome: General Health Status (SF-36)
Description: The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) was used to assess general health status. The SF-36 results are summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). The score for PCS and MCS is between 0 and 100, with higher scores denoting better quality of life.
Time Frame: 24 month after operation
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
Scores on a scale
  Physical Component Summary (PCS) Score at baseline | 27.0 (7.9) | 26.6 (4.7) | 27.0 (3.7) | 24.0 (1.5)
  Physical Component Summary (PCS) Score at 24 month | 44.7 (12.1) | 44.4 (11.8) | 45.2 (12.6) | 46.6 (11.3)
  PCS Score Change at 24 month from baseline | 17.2 (12) | 17.5 (12.4) | 18.1 (11.6) | 22.6 (9.8)
  Mental Component Summary (MCS) Score at baseline | 51.7 (9.2) | 49.7 (10.5) | 46.0 (10.7) | 59.9 (4.2)
  Mental Component Summary (MCS) Score at 24 month | 54.9 (8.8) | 56.7 (9.3) | 55.4 (2.8) | 53.9 (4.1)
  MCS Score Change at 24 month from baseline | 3.6 (9.3) | 2.7 (6.7) | 9.4 (9.2) | -6.0 (0.1)

10. Secondary Outcome: Success Rate of SF-36 Health Survey
Description: Success rate of SF-36 Health Survey include two components: the success rate of a physical component summary (PCS) and the success rate of a mental component summary (MCS). The success rates of SF-36 PCS and MCS for DIAM Device vs. Single-Level Posterior Decompression were defined as: (Post Score - Pre Score) / Pre Score>= 20%. The success rates of SF-36 PCS and MCS for DIAM vs. Posterolateral Interbody Fusion were defined as: Post Score - Pre Score >= 0.
Time Frame: 24 month after operation
Measure: Number; unit: percentage of participants
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 13 | 8 | 4 | 2
percentage of participants
  Success Rate of PCS | 76.9 | 75.0 | 100.0 | 100.0
  Success Rate of MCS | 30.8 | 12.5 | 100.0 | 0.0

11. Secondary Outcome: Operative Time
Time Frame: at the time of operation
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 14 | 12 | 4 | 2
hrs | 1.8 (0.7) | 1.1 (0.6) | 1.2 (0.5) | 2.4 (0.9)

12. Secondary Outcome: Blood Loss
Time Frame: At the time of operation
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 14 | 12 | 4 | 2
ml | 82.5 (68.6) | 77.9 (108.9) | 57.5 (29.9) | 155.0 (63.6)

13. Secondary Outcome: Hospital Stay
Time Frame: At the time of discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Number analyzed (Participants) | 14 | 12 | 4 | 2
days | 1.4 (0.9) | 1.6 (1.0) | 2.0 (1.2) | 3.5 (0.7)

ADVERSE EVENTS:
Time Frame: 24 month
Arm/Group | DIAM Group1 | Single-Level Posterior Decompression | DIAM Group2 | Posterolateral Interbody Fusion
Serious Adverse Events (participants affected / at risk) | 5/14 | 7/12 | 1/4 | 1/2
Other Adverse Events (participants affected / at risk) | 12/14 | 11/12 | 4/4 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DIAM Group1 (N=14) | Single-Level Posterior Decompression (N=12) | DIAM Group2 (N=4) | Posterolateral Interbody Fusion (N=2)
Accidental Injury/ Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiovascular (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cervical spine event (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dural injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal-other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision-related (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Low extremity not of back etiology (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurological (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Other (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal event at target level (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Upper extremity pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urogenital (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DIAM Group1 (N=14) | Single-Level Posterior Decompression (N=12) | DIAM Group2 (N=4) | Posterolateral Interbody Fusion (N=2)
Accidental injury / muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back and/or leg pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Cadiovascular (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dural injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elevated temperature without infection (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hematological (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision-related (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lower extremity not of back etiology (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (3) | 1 (1) | 1 (1)
Neck and arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurological (Nervous system disorders) | 2 (5) | 3 (6) | 1 (2) | 0 (0)
Other (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Other pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Spinal event at other lumbar level (s) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Spinal event at target level (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0)
Trauma (Injury, poisoning and procedural complications) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Upper extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Urogenital (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Studies terminated before full cohort of participants were enrolled. Data and adverse events presented are through 24 months of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must provide the sponsor a copy of the results communication ninety (90) days prior to submission or disclosure. The sponsor shall not censor the results communication beyond the protection of confidential information. Investigator agrees to delete confidential information prior to any submission, publication, presentation or other disclosure. The sponsor can embargo results communications up to sixty (60) days.